CLINICAL TRIAL: NCT07167810
Title: Innovative Approaches to Chest Wall Reconstruction: A Comparative Study of Rigid and Flexible Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Zeeshan Sarwar, Principle Investigator, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB/2025/1542/SIMS
Record Dates: First submitted 2025-09-03; First posted 2025-09-11 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Chest Wall Tumor
Keywords: resection of chest wall; chest wall reconstruction; bone cement; sternal steel wires
MeSH Terms: interventions — Bone Cements

STUDY DESIGN:
Intervention Model Description: This study was a parallel retrospective comparative cohort study conducted at the Thoracic Surgery Unit of Services Hospital, Lahore. The retrospective component included patients who have previously undergone chest wall reconstruction using either PMMA bone cement or No. 05 twisted stainless steel wires.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bone Cement Group (Experimental): participants undergoing chest wall reconstruction using polymethyl methacrylate bone cement were included in this group
  Interventions: Procedure: bone cement
- Steel Wire Group (Experimental): Participants undergoing chest wall reconstruction using no 5 sternal steel wires were included in this group.
  Interventions: Procedure: steel wires

INTERVENTIONS:
Procedure: bone cement — chest wall reconstruction using polymethyl methacrylate PMMA bone cement
  Arms: Bone Cement Group
Procedure: steel wires — chest wall reconstruction using no 05 stainless sternal steel wires
  Arms: Steel Wire Group

SUMMARY:
Chest wall resections, often performed for tumors, infections, or trauma, result in significant defects that require reconstruction to restore structural integrity and functionality. The chest wall, a complex dynamic structure composed of both rigid and soft tissues, plays a vital role in protecting thoracic organs and maintaining the mechanics of respiration. Reconstruction following chest wall resection is critical not only to achieve defect closure but also to preserve respiratory mechanics and minimize postoperative complications. The primary goals include providing structural support, ensuring stability, and achieving soft tissue coverage while maintaining chest wall flexibility and minimizing pain. the main objectives of this study is to compare the postoperative pain control and recovery outcomes between chest wall reconstruction using PMMA bone cement and twisted stainless steel wires in patients undergoing chest wall reconstruction and to evaluate the impact of chest wall reconstruction with steel wires versus PMMA on chest wall recoil.

DETAILED DESCRIPTION:
Various materials and techniques have been employed for chest wall reconstruction, focusing on both soft and rigid defect coverage. Traditional approaches often involve synthetic materials, including mesh, titanium plates, and polymethyl methacrylate (PMMA) bone cement. PMMA, widely known as bone cement, has been a cornerstone material due to its significant compressive strength and ease of application. However, it possesses notable drawbacks, including low tensile strength, lack of adhesive properties, and complications arising from direct exposure to the medullary cavity, such as thermal necrosis, infection, and chronic pain. Studies have also highlighted the static nature of PMMA, which can compromise chest wall dynamics and contribute to suboptimal respiratory outcomes. Furthermore, PMMA is relatively expensive, making it less accessible in resource-constrained settings like Pakistan, where socioeconomic challenges often dictate treatment choices.

In contrast, the use of twisted stainless steel wires (No. 05) for chest wall reconstruction offers a cost-effective and practical alternative. Steel wires provide robust structural support, allow dynamic movement of the chest wall during respiration, and are associated with improved postoperative pain control. Unlike PMMA, which forms a rigid and static patch, steel wires enable better chest wall recoil, which is crucial for maintaining normal respiratory mechanics. Additionally, studies suggest that the use of steel wires reduces the incidence of chronic pain, as they do not involve direct exposure to synthetic materials that could irritate surrounding tissues or provoke inflammatory responses. The affordability and simplicity of steel wire-based reconstruction make it particularly suitable for underserved populations in Pakistan, where healthcare resources are limited, and the majority of patients cannot afford expensive surgical materials.

Chest wall reconstruction techniques that aim to replicate the rib cage's normal anatomy and function have shown promise in improving patient outcomes. Recent innovations, such as neoribs constructed with PMMA, attempt to restore the rib structure and mechanics. However, while effective in achieving structural stability, these techniques often fail to replicate the chest wall's dynamic behavior due to the rigid nature of the material. In contrast, the flexibility and adaptability of steel wires make them an attractive alternative, especially in low-resource settings. Comparative studies have shown that patients reconstructed with steel wires experience less postoperative pain, faster recovery, and better respiratory mechanics than those reconstructed with PMMA.

This study, to be conducted at the Thoracic Surgery Unit of Services Hospital, Lahore, aims to compare the outcomes of chest wall reconstruction using PMMA bone cement versus No. 05 twisted steel wires. The focus will be on evaluating postoperative pain control and chest wall recoil during respiration. Services Hospital, as a tertiary care center and referral unit, manages a significant caseload of thoracic surgeries and serves a predominantly low-income population, making it an ideal setting for this research. By addressing the unique challenges faced by this population and leveraging the available resources, this study seeks to provide evidence-based recommendations for optimizing chest wall reconstruction techniques. The findings are expected to have significant implications for improving patient outcomes and reducing healthcare costs in similar resource-limited settings.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing chest wall resection due to tumors, infections, or trauma.
* Adults aged more than 12 years.
* Patients who provide written informed consent.

Exclusion Criteria:

* Patients with contraindications to surgery.
* Patients with pre-existing chest wall deformities or severe chronic respiratory diseases.
* Patients who undergo reoperation or develop intraoperative complications affecting the chest wall reconstruction.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
post-operative pain | post-operative day 01, day 3 and day 07
  Pain will be assessed using a Visual Analogue Scale (VAS, 0-10 cm), where 0 = no pain and 10 = worst imaginable pain. Assessments will be performed at rest and during deep inspiration/cough. Scores will be collected by trained nursing staff once daily. The primary analysis will report mean VAS score at each time point (with SD).
Chest Wall integrity | day 30 after surgery
  Radiological evaluation, X-ray will be conducted 1 month post-surgery to assess rib alignment and chest wall integrity.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Shoaib Nabi, Principal Investigator — Services Hospital, Lahore
Locations (1):
- Services Institute of Medical Sciences (SIMS), Services Hospital Lahore, Lahore, Punjab Province, Pakistan